CLINICAL TRIAL: NCT00838474
Title: The Effect of Music by Mozart on Energy Expenditure in Growing Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dror Mandel, MD, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 07-346
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2009-02-06 (Estimated); Status verified 2009-02

CONDITIONS: Preterm Infants
Keywords: metabolic rate; music; preterm infants; energy expenditure; NIDCA
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- music therapy (Other): Each infant was randomized to receive music therapy or no music over 2 consecutive days
  Interventions: Other: music

INTERVENTIONS:
Other: music — Each infant was randomized to receive music therapy or no music over 2 consecutive days

SUMMARY:
Music has been consistently shown to reduce stress and increase weight gain in premature infants. The mechanism of this presumed improved metabolic efficiency is unknown. We aim to test the hypothesis that music by Mozart reduces energy expenditure in growing healthy preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* appropriate weight for gestational age
* postmenstrual age of 30-37 weeks
* gavage fed
* tolerating full enteral feedings without significant gastric residuals (>5% of total feed)
* no electrolyte imbalance

Exclusion Criteria:

* congenital anomalies
* dysmorphism
* intracranial hemorrhage of any grade
* periventricular leukomalacia
* necrotizing enterocolitis
* supplemental oxygen requirements by 28 days of age or by 36 weeks of postmenstrual age and at least 1 week prior to measurement
* active infection
* patent ductus arteriosus
* apnea of prematurity

Max Age: 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Energy Expenditure (EE) | during measurment of EE

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neonatology, Tel Aviv Medcil Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Lubetzky R, Mimouni FB, Dollberg S, Reifen R, Ashbel G, Mandel D. Effect of music by Mozart on energy expenditure in growing preterm infants. Pediatrics. 2010 Jan;125(1):e24-8. doi: 10.1542/peds.2009-0990. Epub 2009 Dec 7. PMID 19969615